CLINICAL TRIAL: NCT05802134
Title: Increased Access to Fruits and Vegetables for DASH Diet Compliance in Immigrant Hispanic/Latinx Individuals With Hypertension
Brief Title: Increased Access to Fruits and Vegetables for Hypertension in Immigrant Hispanic/Latinx Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Catherine University (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1744
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
Keywords: carotenoids; cardiovascular disease; medically-tailored food kit; Hispanic/Latinx
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fruit; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruit and Vegetable recipient (Experimental): For 4 weeks, the individuals will receive supplemental, culturally-appropriate fruits and vegetables (to achieve 8-10 servings per day) supported by intensive education for chronic disease management.
  Interventions: Dietary Supplement: Fruit and vegetable supplement; Behavioral: Dietary and chronic disease management education

INTERVENTIONS:
Dietary Supplement: Fruit and vegetable supplement — Weekly food kits including culturally-appropriate fruits and vegetables (to achieve 8-10 servings per day) and staple items to support DASH diet compliance
Behavioral: Dietary and chronic disease management education — Intensive education for chronic disease management: participants will receive education on hypertension management, which will include an interprofessional health appointment with a medical professional to discuss medication compliance, and resources from an occupational therapist for chronic disease management strategies, and 2 nutrition appointments with a Registered Dietitian regarding the DASH Diet (initial education and follow-up at 2 weeks)

SUMMARY:
The goal of this observational study is to learn about the effect improved access to culturally-appropriate fruits/vegetables has on cardiometabolic markers, specifically systolic blood pressure and markers of adiposity in immigrant Hispanic/Latinx individuals with hypertension and obesity. The secondary aim is to determine compliance to the increased F/V intake recommended by the Dietary Approaches to Stop Hypertension (DASH) Diet by assessing changes in skin carotenoid status. The main question it aims to answer is whether consuming 8-10 servings of culturally-appropriate, carotenoid-containing F/V daily for 4 weeks to meet the requirements of the DASH Diet supported by diet and lifestyle education will result in reductions in systolic BP and decreased markers of adiposity (body weight, Body Mass Index, and waist circumference).

DETAILED DESCRIPTION:
This study will utilize a phased, mixed methods approach including a literature review to inform a patient/provider survey, individual patient interviews to better understand how to develop a medically-tailored foods box for the patient population with hypertension, and an open observational study.

The proposed study will be conducted at a St. Mary's Health Clinics site in the Twin Cities metro, which includes access to the required equipment, a space to collect required measures, and designated patient rooms for participant privacy. Obese (BMI >30 kg/m2) men and women (ages 18+) diagnosed with hypertension will be recruited via flyers, email, and mail from St. Mary's Health Clinics for an open observational study. For 4 weeks, the individuals will receive supplemental, culturally-appropriate fruits and vegetables (to achieve 8-10 servings per day) supported by intensive education for chronic disease management. To address social determinants of health surrounding fruit and vegetable access, food will be provided for the patient and family members, if the participant indicates a need.

Participants will receive supplemental fruits and vegetables high in carotenoids and staple items that are promoted on a DASH Diet, with encouragement and support to consume the fruits and vegetables via recipes, samples, and weekly text/call check-ins to support utilization. Compliance will be measured via non-invasive skin carotenoid status using a Veggiemeter. Boxes will be distributed from a central site, similar to the medication pick-up structure St. Mary's Health Clinics patients are familiar with or will be delivered to the patient's preferred address, if access to the clinic is a barrier. All enrolled participants will receive education on hypertension management, which will include an interprofessional health appointment with a medical professional to discuss medication compliance, and resources from an occupational therapist for chronic disease management strategies, and 2 nutrition appointments with a Registered Dietitian regarding the DASH Diet (initial education and follow-up at 2 weeks). The interprofessional education provided is intended to yield in higher compliance to dietary changes and adherence to medication regimen. All materials and appointments will be available in Spanish and English. There will be an interpreter available for all medical appointments, as 85% of patients are non-English speaking.

All participants will be screened to ensure eligibility. Screening will include: a demographic (age, gender, race/ethnicity, smoking status, family size, and primary food preparer in the household) and medical history questionnaire to determine comorbidities. The National Cancer Institute's 19-item F/V screener will be utilized to determine regular consumption of F/V for the participant and the family, if applicable. Exclusions will be made for individuals that are taking insulin to manage diabetes mellitus, smokers, and those with a BMI <30 kg/m2. At baseline (day 0) and Day 28, cardiometabolic markers (height, weight, BP, waist circumference, and skin carotenoid status) will be collected. BP will be measured by trained professionals using random- zero sphygmomanometers while sitting down after a 5-minute rest period. Two measures will be collected and averaged. Carotenoid status will be assessed via non-invasive skin spectrometry using a VeggieMeter (Longevity Link Corporation, UT). The quantity of F/V provided in the supplemental box to achieve 8-10 servings daily will be determined during the screening.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Hispanic/Latinx individuals
* patients at the St. Mary's Health Clinic
* hypertension diagnosis
* obese (BMI >30 kg/m2)

Exclusion Criteria:

* current smokers
* individuals taking insulin to manage diabetes mellitus
* individuals with a BMI <30 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 1 month
  measure the change in systolic blood pressure while following DASH Diet fruit and vegetable requirements

SECONDARY OUTCOMES:
Diastolic Blood Pressure | 1 month
  measure the change in diastolic blood pressure while following DASH Diet fruit and vegetable requirements
Skin carotenoid status | 1 month
  measure the change in serum carotenoid status using skin spectrometry while following DASH Diet fruit and vegetable requirements

CONTACTS AND LOCATIONS:
Overall Officials: Ambria C Crusan, PhD, Principal Investigator — St. Catherine University
Locations (5):
- United States (5):
  - M Health Fairview Clinic, Apple Valley, Minnesota
  - Church of St. William, Fridley, Minnesota
  - Park Avenue United Methodist Church, Minneapolis, Minnesota
  - St. Catherine University, Saint Paul, Minnesota
  - St. Matthew's Parish Center, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Institute of Health. Eating At America's Table Study Quick Food Scan. Published online 2000. https://snaped.fns.usda.gov/library/materials/national-cancer-institute-nci-fruit-vegetable-intake-screeners-eating-americas-0
- [Background] Chiu S, Bergeron N, Williams PT, Bray GA, Sutherland B, Krauss RM. Comparison of the DASH (Dietary Approaches to Stop Hypertension) diet and a higher-fat DASH diet on blood pressure and lipids and lipoproteins: a randomized controlled trial. Am J Clin Nutr. 2016 Feb;103(2):341-7. doi: 10.3945/ajcn.115.123281. Epub 2015 Dec 30. PMID 26718414
- [Background] Di Noia J, Gellermann W. Use of the Spectroscopy-Based Veggie Meter(R) to Objectively Assess Fruit and Vegetable Intake in Low-Income Adults. Nutrients. 2021 Jun 30;13(7):2270. doi: 10.3390/nu13072270. PMID 34209048
- [Background] Toh DWK, Sutanto CN, Loh WW, Lee WY, Yao Y, Ong CN, Kim JE. Skin carotenoids status as a potential surrogate marker for cardiovascular disease risk determination in middle-aged and older adults. Nutr Metab Cardiovasc Dis. 2021 Feb 8;31(2):592-601. doi: 10.1016/j.numecd.2020.10.016. Epub 2020 Oct 26. PMID 33358716
- [Background] USDA. Food Security Survey Module: Six-Item Short Form. Published 2012. https://snaped.fns.usda.gov/library/materials/food-security-survey-module-six-item-short-form
- [Background] Chiavaroli L, Viguiliouk E, Nishi SK, Blanco Mejia S, Rahelic D, Kahleova H, Salas-Salvado J, Kendall CW, Sievenpiper JL. DASH Dietary Pattern and Cardiometabolic Outcomes: An Umbrella Review of Systematic Reviews and Meta-Analyses. Nutrients. 2019 Feb 5;11(2):338. doi: 10.3390/nu11020338. PMID 30764511
- [Background] Jahns L, Johnson LK, Mayne ST, Cartmel B, Picklo MJ Sr, Ermakov IV, Gellermann W, Whigham LD. Skin and plasma carotenoid response to a provided intervention diet high in vegetables and fruit: uptake and depletion kinetics. Am J Clin Nutr. 2014 Sep;100(3):930-7. doi: 10.3945/ajcn.114.086900. Epub 2014 Jul 9. PMID 25008856
- [Background] Juraschek SP, Woodward M, Sacks FM, Carey VJ, Miller ER 3rd, Appel LJ. Time Course of Change in Blood Pressure From Sodium Reduction and the DASH Diet. Hypertension. 2017 Nov;70(5):923-929. doi: 10.1161/HYPERTENSIONAHA.117.10017. PMID 28993451
- [Derived] Crusan A, Roozen KL, Godoy-Henderson C, Evans A, Reeves K. Developing and evaluating a culturally-appropriate food kit for increased access to fruits and vegetables and DASH eating plan alignment in immigrant Hispanic/Latine individuals with hypertension: a pilot study. BMC Nutr. 2025 May 16;11(1):97. doi: 10.1186/s40795-025-01089-z. PMID 40380253
- See also: DASH Eating Plan — https://www.nhlbi.nih.gov/education/dash-eating-plan
- See also: NIMHD Research Framework — https://www.nimhd.nih.gov/about/overview/research-framework/nimhd-framework.html